CLINICAL TRIAL: NCT05197686
Title: Early-initiated High Flow Oxygen Therapy vs Conventional Oxygen Therapy Among Patients With ARDS in the Course of SARS-CoV2 Pneumonia: Prognosis and Impact on the Respiratory and Cardiovascular Systems.
Brief Title: Early-initiated High Flow Oxygen Therapy vs Conventional Oxygen Therapy Among Patients With ARDS in the Course of SARS-CoV2 Pneumonia.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KB-0012/58/2021
Record Dates: First submitted 2022-01-18; First posted 2022-01-19 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Corona Virus Infection; ARDS Due to Disease Caused by Severe Acute Respiratory Syndrome Coronavirus 2; Oxygen Deficiency
Keywords: SARS-CoV2, COVID-19, HFNC, COT, Oxygen therapy.
MeSH Terms: conditions — Coronavirus Infections; Hypoxia; COVID-19 | interventions — Masks

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Groups are designed by web randomizer.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HFNC (Experimental)
  Interventions: Device: Oxygen theraphy with high flow nasal cannule
- COT (Active Comparator)
  Interventions: Device: Oxygen theraphy with mask with reservoir

INTERVENTIONS:
Device: Oxygen theraphy with high flow nasal cannule — Oxygen theraphy with high flow nasal cannule
  Arms: HFNC
Device: Oxygen theraphy with mask with reservoir — Oxygen theraphy with mask with reservoir
  Arms: COT

SUMMARY:
The aim of the study is to compare two methods of oxygen therapy in patients with acute respiratory distress syndrome in the course of SARS-CoV2 pneumonia. The initial method of oxygen supply during coronavirus pneumonia is conventional oxygen therapy using a face mask or nasal cannula. However, there have been reports in the literature that early initiation of high-flow oxygen therapy with a nasal cannula is associated with better prognosis. The study we perform is intended to provide reliable evidence for confirmation this hypothesis.

ELIGIBILITY:
Inclusion Criteria:

1. The diagnosis of a current SARS-CoV2 infection (confirmed RT-PCR test or antigen test [allowed in Poland, with sensitivity ≥90 and specificity ≥97]);
2. Hospitalization in the Oxygen Sector of the Temporary Hospital in Szczecin;
3. Pneumonia during SARS-CoV2 infection;
4. ARDS (PaO 2 / FiO 2 ratio ≤300);
5. Oxygen flow 8-12 l / min on mask with reservoir and ≤ 60 mmHg paO2 and / or SpO2 < 92%;
6. TNo current indications for treatment in the ICU;
7. Permisson of the patient.

Exclusion Criteria:

1. Probable lack of cooperation with patient;
2. Severe Disease disease, eg generalized neoplastic disease;
3. Concomitant pulmonary diseases (eg, fibrosis lungs);
4. Respiratory acidosis - pH <7.3 with pCO2> 50 mmHg;
5. Disturbances of consciousness - GCS < 12;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-01-18 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Lower mortality in HFNC group | 6 months
Lower percent of intubation in HFNC group | 6 months
Shorter time of hospitalization in HFNC group | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Oxygen Therapy Sector of Temporary Hospital, Szczecin, West Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Baker KF, Hanrath AT, Schim van der Loeff I, Kay LJ, Back J, Duncan CJ. National Early Warning Score 2 (NEWS2) to identify inpatient COVID-19 deterioration: a retrospective analysis. Clin Med (Lond). 2021 Mar;21(2):84-89. doi: 10.7861/clinmed.2020-0688. Epub 2021 Feb 5. PMID 33547065
- [Background] Sayan I, Altinay M, Cinar AS, Turk HS, Peker N, Sahin K, Coskun N, Demir GD. Impact of HFNC application on mortality and intensive care length of stay in acute respiratory failure secondary to COVID-19 pneumonia. Heart Lung. 2021 May-Jun;50(3):425-429. doi: 10.1016/j.hrtlng.2021.02.009. Epub 2021 Feb 10. PMID 33621840
- [Background] Xu Q, Wang T, Qin X, Jie Y, Zha L, Lu W. Early awake prone position combined with high-flow nasal oxygen therapy in severe COVID-19: a case series. Crit Care. 2020 May 24;24(1):250. doi: 10.1186/s13054-020-02991-7. No abstract available. PMID 32448330
- [Background] Vianello A, Arcaro G, Molena B, Turato C, Sukthi A, Guarnieri G, Lugato F, Senna G, Navalesi P. High-flow nasal cannula oxygen therapy to treat patients with hypoxemic acute respiratory failure consequent to SARS-CoV-2 infection. Thorax. 2020 Nov;75(11):998-1000. doi: 10.1136/thoraxjnl-2020-214993. Epub 2020 Jul 23. PMID 32703883
- [Background] Rorat M, Szymanski W, Jurek T, Karczewski M, Zelig J, Simon K. When Conventional Oxygen Therapy Fails-The Effectiveness of High-Flow Nasal Oxygen Therapy in Patients with Respiratory Failure in the Course of COVID-19. J Clin Med. 2021 Oct 16;10(20):4751. doi: 10.3390/jcm10204751. PMID 34682874